CLINICAL TRIAL: NCT04854655
Title: Evaluation of Calcium and Phosphate Releasing Hybrid Restorative Material and Fluoride Releasing Hybrid Restorative Material Versus the Conventional Resin Composite in Proximal Carious Lesions Over One Year Follow-up Using USPHS Criteria
Brief Title: Evaluation of Ion Releasing Hybrid Restorative Material
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nouran Osama El-Sayed Ahmed Abou El-Nour, Resident at Faculty of Dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1994
Record Dates: First submitted 2021-04-20; First posted 2021-04-22 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Conventional resin composite
  Interventions: Other: Conventional resin composite
- Intervention 1 (Experimental): Activa Presto
  Interventions: Other: Activa Presto
- Intervention 2 (Experimental): Giomer
  Interventions: Other: Giomer

INTERVENTIONS:
Other: Conventional resin composite — nanofilled resin composite
  Arms: Control
Other: Activa Presto — calcium and phosphate hybrid material
  Arms: Intervention 1
Other: Giomer — fluoride releasing hybrid material
  Arms: Intervention 2

SUMMARY:
Esthetic and mechanical evaluation of calcium and phosphate releasing hybrid restorative material and fluoride releasing hybrid restorative material versus the conventional nanofilled resin composite in proximal carious lesions over 1 year follow-up according to the USPHS criteria.

DETAILED DESCRIPTION:
3 groups of 45 patients will receive class II restorations by using calcium and phosphate releasing hybrid restorative material (Activa Presto), fluoride releasing hybrid restorative material (Giomer), and conventional nanofilled resin composite. Then these restorations evaluated at 24 hours after placement, 1 month, 3 months, 6 months and 12 months according the modified USPHS criteria in terms of fracture, marginal adaptation, retention, anatomic form, marginal discoloration, surface texture, and color match.

ELIGIBILITY:
Inclusion Criteria:

* Patient-related criteria:

  * Patients consulting in one of the outpatient clinics listed above.
  * Patients can tolerate necessary restorative procedures.
  * Provide informed consent.
  * Patients accept the one year follow-up period.
  * Patients are within middle age group (25-40years).
  * Cooperative patients.
  * Patients don't have any medically compromised conditions.

Tooth related criteria:

* Teeth with primary proximal carious lesions in posterior teeth with no pulpal involvement.
* Teeth should have contact with the adjacent teeth.
* Teeth are vital according to pulp-sensitivity tests.
* No active gingival or periodontal conditions.

Exclusion Criteria:

* • Medically compromised patients, as they will not be able to attend multiple appointments or may require special management.

  * Pregnant women; as radiographs are prohibited.
  * Allergic Patients to any of the restorative materials, including anesthetics.
  * Uncooperative patients will not follow the instructions or attend the appointments.

Tooth related criteria:

* Retained deciduous teeth; as the research is targeting only permanent teeth.
* Teeth with previous restorations, which may add another variable to the study (type of old restorative material, extent of recurrent caries).
* Spontaneous pain or prolonged pain after sensitivity tests (cold and electrical tests) indicating irreversible pulpitis.
* Negative sensitivity tests, periapical radiolucencies, and sensitivity to axial or lateral percussion indicating pulp necrosis.
* Teeth presenting external or internal resorption, with adverse pulpal reactions which may affect the outcome of the study.
* Teeth with cervical caries; which can't be evaluated on periapical radiographs.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-10-10 (Estimated); Primary Completion 2022-10-10 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Mechanical evaluation according to USPHS criteria | 1 year
  Fracture, Retention, Marginal adaptation, Anatomic form, and Surface roughness

SECONDARY OUTCOMES:
: Esthetic evaluation according to USPHS criteria. : Esthetic evaluation according to USPHS criteria. Esthetic evaluation according to USPHS criteria | 1 year
  Color match, marginal discoloration, and restoration color stability